CLINICAL TRIAL: NCT03156491
Title: The Maternal-embryo Interaction and Its Role in the Etiology of Recurrent Miscarriages
Brief Title: Maternal Embryo Interaction in Recurrent Miscarriages
Acronym: MEER
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Bart CJM Fauser, Professor, UMC Utrecht
Other Study IDs: MEER-study; METC (Registry Identifier: 09-408/C); CCMO (Registry Identifier: NL30143.000.09)
Record Dates: First submitted 2010-04-01; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Recurrent Miscarriages
Keywords: recurrent miscarriages (RM); recurrent pregnancy loss (RPL); fetal-maternal interface; decidualization; co-culture; implantation; immune regulation
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — endometrial biopsies and peripheral blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Recurrent miscarriage group: Women with unexplained recurrent miscarriages (three or more first trimester miscarriages).
- Control group: Proven fertile women (at least 1 successful pregnancy and no more than 1 miscarriage).

SUMMARY:
Background of the study:

The etiology of recurrent miscarriage (RM, defined as three or more consecutive miscarriages without any proven maternal or fetal cause), remains undiagnosed in more than 50% of cases. In these cases it is generally considered that a disturbance in the normal mother-embryo interactions is a causal factor. This disturbance may be based on a dysregulation of embryo invasiveness and/or decidual acceptance (e.g. altered decidualization; endometrial changes in preparation for the acceptance of a putative pregnancy). Moreover, dysfunctional maternal immune regulatory natural killer (NK) cells, implicated in tolerance induction and trophoblast invasion,may also underlie the occurrence of RM. The Selection Failure hypothesis for RM suggests that super-receptive endometrium (possibly due to increased embryo invasiveness and/or decidual acceptance and/or dysregulated immune cell function) may allow 'poor quality' embryos to implant and present as a clinical pregnancy before miscarrying. Fundamental knowledge on mechanisms of embryo implantation, decidual function and maternal immune reactivity in successful pregnancies has accumulated over the past 5 years. This study aims to investigate whether dysregulation of (one of) these mechanisms may underlie RM.

Objective of the study:

To test The Selection Failure hypothesis by assessing A) the degree of embryo invasiveness and decidual acceptance (the quality of decidualization, endometrium-embryo communication and endometrial stromal cell (ESC) migration) and B) the angiogenic capacity of decidual NK (dNK) cells, in order to elucidate the pattern of the mother-embryo equilibrium in women with RM.

ELIGIBILITY:
Inclusion Criteria:

1. Women with unexplained recurrent miscarriages (three or more first trimester miscarriages).
2. Proven fertile women (at least 1 successful pregnancy and no more than 1 miscarriage).
3. Age 18 - 40 years.
4. Willing and able to give informed consent.

Exclusion Criteria:

1. Any identifiable causes of recurrent miscarriages; antiphospholipid syndrome (lupus anticoagulant and/or anticardiolipin antibodies [IgG or IgM]), other recognised thrombophilic conditions (testing according to usual clinic practice), intrauterine abnormalities (as assessed by ultrasound, hysterosonography, hysterosalpingogram or hysteroscopy), submucous fibroids and tests initiated only if clinically indicated such as tests for diabetes, thyroid disease and SLE
2. Undergoing treatment (hormonal)
3. Women using oral contraception or having an intra uterine device.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recurrent miscarriage group: primary care clinic Control group: primary care clinic/community sample
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Embryo survival on decidualized ESCs of RM patients or fertile controls (Embryo survival as an indirect measure of embryo invasiveness) | 2 years
  Embryo survival as an indirect measure of embryo invasiveness

CONTACTS AND LOCATIONS:
Overall Officials: Cobi J Heijnen, Prof. dr., Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided